CLINICAL TRIAL: NCT02641145
Title: Molecular Imaging of Primary Amyloid Cardiomyopathy
Acronym: MICA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Sharmila Dorbala, Director, Nuclear Cardiology, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P002477; 1R01HL130563-01A1 (NIH)
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Amyloidosis, Primary; Cardiomyopathy
Keywords: amyloidosis; F-18 florbetapir; Positron emission tomography; cardiac magnetic resonance imaging
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Cardiomyopathies; Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Active AL cardiac amyloidosis (Experimental): 75 individuals with light chain systemic amyloidosis with active plasma cell dyscrasia and cardiac involvement will undergo a research F-18 florbetapir PET, C-11 acetate PET, and MRI of blood of the heart, as well as the heavy metal analysis of the blood at baseline, 6 months and 12 months after initiation of chemotherapy. 25 of these individuals will also undergo a N-13 ammonia PET scan of the heart following supine bicycle stress at baseline and at 6 months after initiation of chemotherapy.
  Interventions: Radiation: F-18 florbetapir/C-11 acetate PET; Device: MRI; Radiation: N-13 ammonia PET
- Remission AL cardiac amyloidosis (Active Comparator): 25 individuals with light chain systemic amyloidosis with cardiac involvement and plasma cell dyscrasia in hematological remission (complete hematological remission or very good partial response-differential free light chain (dFLC)<40 mg/dL for > 1 year prior to enrollment) will undergo a research F-18 florbetapir PET, C-11 acetate PET, and MRI scan of the heart as well as a heavy metal analysis of the blood at baseline.
  Interventions: Radiation: F-18 florbetapir/C-11 acetate PET; Device: MRI
- Active AL Pre-CMP (Experimental): 36 individuals with light chain systemic amyloidosis with active plasma cell dyscrasia and without cardiac involvement will undergo a research F-18 florbetapir PET, C-11 acetate PET, and MRI of the heart, as well as a heavy metal analysis of the blood at baseline. At 6 months they will undergo a research MRI of the heart and at 12 months they will have a clinical follow up. Subjects with contraindications to Cardiac MRI or gadolinium contrast may still be eligible for study participation.
  Interventions: Radiation: F-18 florbetapir/C-11 acetate PET; Device: MRI
- Multiple Myeloma Controls (No Intervention): 25 individuals with diagnosis of multiple myeloma without concomitant amyloidosis by standard criteria will undergo urine and blood testing only.
- Heart Failure (Experimental): 10 individuals with diagnosis of heart failure without amyloidosis by standard criteria will undergo a research F-18 florbetapir PET, C-11 acetate PET, and MRI of the heart, as well as a heavy metal analysis of the blood at baseline..
  Interventions: Radiation: F-18 florbetapir/C-11 acetate PET; Device: MRI

INTERVENTIONS:
Radiation: F-18 florbetapir/C-11 acetate PET — F-18 florbetapir PET scan, C-11 acetate PET scan
  Arms: Active AL Pre-CMP; Active AL cardiac amyloidosis; Heart Failure; Remission AL cardiac amyloidosis
Device: MRI — Cardiac MRI with gadolinium contrast.
  Arms: Active AL Pre-CMP; Active AL cardiac amyloidosis; Heart Failure; Remission AL cardiac amyloidosis
Radiation: N-13 ammonia PET — N-13 ammonia PET scan following supine bicycle stress.
  Arms: Active AL cardiac amyloidosis

SUMMARY:
Cardiac amyloidosis is a major cause of early treatment-related death and poor overall survival in individuals with systemic light chain amyloidosis. This project will develop a novel approach to visualize cardiac amyloid deposits using advanced imaging methods. The long-term goal of this work is to identify the mechanisms of cardiac dysfunction, in order to guide the development of novel life-saving treatments.

DETAILED DESCRIPTION:
Primary light chain amyloidosis (AL) is the most common systemic amyloidosis, resulting from a plasma cell dyscrasia, a hematological malignancy. It causes a restrictive cardiomyopathy (AL-CMP) in over 70% of individuals. AL-CMP is as lethal as stage 4 lung cancer and more lethal than any other form of restrictive heart disease; if untreated, the mortality rate is 50% within 18 months. Moreover, myocardial dysfunction, the hallmark of AL-CMP, significantly increases early treatment related mortality, predominantly cardiovascular death, and is a powerful predictor of poor long-term survival. Two potentially treatable mechanisms underlie myocardial dysfunction-mechanical effects of amyloid and toxic effects from circulating light chain/ amyloid interactions-and predispose to heart failure, arrhythmias, and sudden death in individuals with AL-CMP. Until now, efforts to determine the mechanisms of AL-CMP have been hampered by a lack of animal models and the limitations of noninvasive techniques to directly image myocardial amyloid. A recent breakthrough, 18F-florbetapir PET/CT, has provided for the first time specific and quantitative imaging of myocardial amyloid including toxic amyloid protofibrils. Furthermore, we propose to investigate three pre-clinically proven pathways of light chain toxicity in humans-myocardial oxidative metabolism, oxidative stress, and coronary microvascular function. Our central hypotheses are that myocardial 18F-florbetapir retention is a biomarker for aggressiveness of AL-CMP and that effective chemotherapy will, by reducing circulating light chains, decrease aggressiveness of AL-CMP and improve oxidative stress, myocardial oxidative metabolism, microvascular function and contractile function, prior to an improvement in myocardial amyloid content. In Aim 1, we will quantify myocardial 18F-florbetapir retention as a marker of aggressive myocardial disease in individuals with AL-CMP and active plasma cell dyscrasia compared to control individuals with AL-CMP and long-term hematological remission. In Aim 2, we propose, using advanced imaging, to assess the effects of light chain reduction due to chemotherapy on myocardial structure, function, and metabolism and define the time course of these changes. Serial ECV and strain imaging by CMR, serum F2-isoprostanes and peroxynitrite levels, myocardial oxidative metabolism (Kmono) and coronary flow reserve by 11C-acetate PET, and 18F-florbetapir imaging will not only intricately characterize the myocardial substrate in AL-CMP, but also identify changes in response to therapy. The proposed studies offer the potential to transform our current understanding of AL-CMP as a restrictive heart disease caused by passive amyloid-related architectural damage to that of a more complex disorder resulting from both passive and aggressive factors. The results of these studies may form the foundation for drug discovery programs to prevent and cure AL-CMP.

Interactions of environmental factors, immunity, and host-related factors likely trigger AL-amyloidosis, but have not yet been explored. Changes in metal ions and gut microbiota may be causal, representing the integrated effects of all these factors, or may be the downstream effect of systemic amyloid deposition in the organ systems. A plethora of recent literature strongly support the role of microbiota in the pathogenesis of several diseases, suggesting that gut microbiota changes with age, influences heart failure (HF) outcomes, and plays a role in the formation of β-amyloid deposits in Alzheimer's disease. Importantly, alterations in lifestyle, diet, prebiotics, probiotics, or phenols and gut microbiota may represent therapeutic and preventative strategies in amyloid disease, but it has not been explored in AL-amyloidosis. We propose to study the role of salivary and gut microbiome in AL amyloidosis.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Diagnosis of light chain amyloidosis by standard criteria (immunofixation of serum and urine, IgG free light chain (FLC) assay, a biopsy of fat pad/ bone marrow, or organ biopsy, followed by typing of the light chain using immunohistochemistry or immunogold assay with confirmation by Mass spectroscopy as needed)

  * For subjects traveling from out of town referred for systemic AL therapy based on clinical evaluation and laboratory testing, but, pending biopsy results, study enrollment and procedures may begin before official confirmation of biopsy results. If biopsy is negative for AL amyloidosis, subject will be considered a screen failure. There will be no more than 10 subjects who fall under this screen failure for the duration of the study.
  * Subjects with localized amyloid deposition and non-systemic AL disease will be eligible for enrollment in group D.
* Willing and able to provide consent
* Additional inclusion criteria for the Remission AL-CMP: Hematological response defined as complete hematological remission or very good partial response-differential free light chain (dFLC)<40 mg/dL for > 1 year prior to enrollment
* Additional inclusion criteria for the Active AL-CMP - exercise: Ability to perform supine bicycle exercise. Enrollment to this arm will stop after 36 subjects complete baseline and 6 months studies.
* Additional inclusion criteria for the Active AL Pre-CMP - Normal left ventricular wall thickness (≤ 12 mm) and normal LVEF (≥55%) on echocardiography within 3 months or increased wall thickness with normal cardiac biomarker levels: not meeting above definition.
* Additional inclusion criteria for Control Multiple Myeloma subjects: diagnosis of multiple myeloma without concomitant amyloidosis by standard criteria
* Additional inclusion criteria for Control Heart Failure subjects: diagnosis of heart failure without amyloidosis by standard criteria
* Additional inclusion criteria for the active AL-CMP: Abnormal TnT 5th generation levels (>9 ng/L: Female, >14 ng/L: Male) or abnormal age appropriate N terminal pro-brain natriuretic peptide, NT-proBNP (abnormal values: <50 years: >450 pg/ml; 50-75 years:>900 pg/ml; >75 years: >1800 pg/ml)

Exclusion Criteria:

* Hemodynamic instability
* Decompensated heart failure (unable to lie flat for 1 hour)
* Concomitant non-ischemic non-amyloid heart disease (valvular heart disease or dilated cardiomyopathy)
* Known obstructive epicardial coronary artery disease with stenosis > 50% in any single territory
* Severe claustrophobia despite use of sedatives
* Presence of MRI contraindications such as metallic implants (pacemaker or ICD) at the time of study enrollment except for Control Heart Failure subjects. Control HF subjects with no devices, or, with strictly MR compatible devices will be eligible to undergo MRI.
* Significant renal dysfunction with estimated glomerular filtration rate < 30 ml/min/m2 within 14 days of each cardiac MRI study. Subjects who develop renal dysfunction over the course of the study, meeting criteria listed above, will be excluded from the cardiac MRI scan except for control HF subjects. These subjects with eGFR < 30 ml/min/1.73 m2 will undergo MRI without gadolinium contrast.
* Subjects on dialysis will be excluded
* Pregnant state. For women in child bearing age, a urine pregnancy test will be performed prior to the PET and the cardiac MRI studies
* Documented allergy to F-18 florbetapir, C-11 acetate or gadolinium.
* Additional exclusion criteria for the active AL-CMP subjects: Subjects unable to return to BWH for 6 and 12 month clinical evaluation
* Additional exclusion criteria for active AL-CMP-exercise subjects: Inability to exercise or return to BWH for C-11 acetate PET/CT at baseline and 6 month clinical evaluations.
* Additional exclusion criteria for active AL Pre-CMP- Inability to return to BWH 12 month clinical evaluation.

Additional exclusion criteria for microbiota study: Documented hypertrophic cardiomyopathy, HIV or chronic viral hepatitis, documented inflammatory bowel disease, systemic antibiotics, antivirals, antifungals or antiparasitic agents within 6 months, unable to mail the stool sample in a timely manner, bowel surgery, colon cancer, received chemotherapy, and pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2016-04-01; Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in F-18 florbetapir myocardial retention index from baseline to 6 months and 12 months | Baseline, 6 and 12 months
  quantitative measure of F-18 florbetapir uptake by the heart muscle
Change in Serum oxidative stress markers from baseline to 6 months and 12 months | Baseline, 6 and 12 months
  serum F-2 isoprostane and peroxynitrite levels
Change in Myocardial oxidative metabolism markers from baseline to 6 months | Baseline and 6 months
  K mono and coronary flow reserve obtained by C-11 acetate PET/CT at rest and stress
Change in Magnetic resonance imaging markers from baseline to 6 months and 12 months | Baseline, 6 and 12 months
  Extracellular volume index, T-1 mapping, late gadolinium enhancement, global strain, left ventricular mass

SECONDARY OUTCOMES:
Change in Myocardial energy efficiency from baseline to 6 months | Baseline and 6 months
  Myocardial energy efficiency, Kmono reserve, will be determined by C-11 acetate PET
Light Chain Toxicity | Baseline
  Study subject urine light chain's will be extracted and infused into zebrafish and isolated cardiomyocytes to study light chain toxicity
Understand the role of gut microbiota and heavy metals in the pathogenesis of AL Amyloidosis | Baseline
  This will be tested using machine learning methods with 16S rRNA sequencing of salivary and stool samples in a 40-patient cohort with AL-amyloidosis compared to healthy controls from the NIH funded human microbiome project (HMP).This will also be used to test if the gut microbiome affects amyloid formation using a transgenic mouse model of AL amyloidosis that expresses the human LC in the gut and develops amyloid in the stomach.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Dorbala, MD, Principal Investigator — Brigham and Women's Hospital (AHA and NIH Studies); Rodney Falk, MD, Principal Investigator — Brigham and Women's Hospital (NIH Study); Ronglih Liao, PhD, Principal Investigator — Stanford School of Medicine (AHA Study)
Locations (1):
- Brigham and Womens' Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not have a plan to share individual participant data with other researchers

REFERENCES:
- [Derived] Benz DC, Clerc OF, Cuddy SAM, Singh V, Kijewski MF, Bianchi G, Yee AJ, Ruberg FL, Jerosch-Herold M, Kwong RY, Di Carli MF, Liao R, Falk RH, Dorbala S. Changes in Myocardial Light Chain Amyloid Burden After Plasma Cell Therapy. JACC Cardiovasc Imaging. 2025 Dec;18(12):1363-1374. doi: 10.1016/j.jcmg.2025.07.017. Epub 2025 Sep 12. PMID 40938234
- [Derived] Clerc OF, Cuddy SAM, Jerosch-Herold M, Benz DC, Katznelson E, Canseco Neri J, Taylor A, Kijewski MF, Bianchi G, Ruberg FL, Di Carli MF, Liao R, Kwong RY, Falk RH, Dorbala S. Myocardial Characteristics, Cardiac Structure, and Cardiac Function in Systemic Light-Chain Amyloidosis. JACC Cardiovasc Imaging. 2024 Nov;17(11):1271-1286. doi: 10.1016/j.jcmg.2024.05.004. Epub 2024 Jul 10. PMID 39001736
- [Derived] Katznelson E, Jerosch-Herold M, Cuddy SAM, Clerc OF, Benz DC, Taylor A, Rao S, Kijewski MF, Liao R, Landau H, Yee AJ, Ruberg FL, Di Carli MF, Falk RH, Kwong RY, Dorbala S. Mechanisms of left ventricular systolic dysfunction in light chain amyloidosis: a multiparametric cardiac MRI study. Front Cardiovasc Med. 2024 May 30;11:1371810. doi: 10.3389/fcvm.2024.1371810. eCollection 2024. PMID 38873265
- [Derived] Cuddy SAM, Jerosch-Herold M, Falk RH, Kijewski MF, Singh V, Ruberg FL, Sanchorawala V, Landau H, Maurer MS, Yee AJ, Bianchi G, Di Carli MF, Liao R, Kwong RY, Dorbala S. Myocardial Composition in Light-Chain Cardiac Amyloidosis More Than 1 Year After Successful Therapy. JACC Cardiovasc Imaging. 2022 Apr;15(4):594-603. doi: 10.1016/j.jcmg.2021.09.032. Epub 2021 Dec 15. PMID 34922860
- [Derived] Cuddy SAM, Bravo PE, Falk RH, El-Sady S, Kijewski MF, Park MA, Ruberg FL, Sanchorawala V, Landau H, Yee AJ, Bianchi G, Di Carli MF, Cheng SC, Jerosch-Herold M, Kwong RY, Liao R, Dorbala S. Improved Quantification of Cardiac Amyloid Burden in Systemic Light Chain Amyloidosis: Redefining Early Disease? JACC Cardiovasc Imaging. 2020 Jun;13(6):1325-1336. doi: 10.1016/j.jcmg.2020.02.025. Epub 2020 May 13. PMID 32417333